CLINICAL TRIAL: NCT07038395
Title: Retrospective Comparative Analysis of Time and Motion Workflow of Femtosecond Laser-assisted Cataract Surgery (FLACS) in Multiple Surgical Settings
Brief Title: Retrospective Analysis of the Time Elements for Different Workflow Scenarios During Femtosecond Laser-assisted Cataract Surgery (FLACS) From the Surgeon, Staff, and Patient Perspectives.
Status: Completed | Type: Observational
Sponsor: LensAR Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: ME-00008-PRO
Record Dates: First submitted 2025-05-20; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Nonsterile feeder room model: Procedures performed in a separate room from the operating room
  Interventions: Device: workflow
- Sterile room model: Procedures performed in a sterile environment
  Interventions: Device: workflow

INTERVENTIONS:
Device: workflow — Placement of the surgical device and its effect on workflow

SUMMARY:
This study involves the retrospecitve review of time stamps during surgery to assess the time efficiencies of different workflow scenarios of femtosecond laser-assisted cataract surgery from the surgeon, staff, and patient perspectives.

Objectives are to identify surgical workflows that may increase surgical efficiency and improve patient, surgeon, and staff satisfaction.

DETAILED DESCRIPTION:
Cataracts are the most common cause of preventable visual impairment. In the United States, the number of people with cataracts is forecasted to double from 24.4 million to about 50 million by the year 20501. By age 80, half of all Americans have a cataract. Recent and ongoing reductions in reimbursement for cataract surgery have fueled an increased need to drive innovation in ways to be more financially efficient. Simultaneously, new technology in the field, especially as it relates to use of the femtosecond laser for portions of lens surgery, can increase challenges in creating an efficient and cost-effective structure for providing care2.

Understanding operating room workflows is crucial for cataract surgeons, as it allows them to improve efficiency, achieve time savings, and realize significant cost savings. By optimizing workflows, surgeons can streamline processes, reduce delays, and expedite surgical procedures, leading to shorter wait times for patients. Moreover, efficient resource utilization, including surgical instruments and equipment, minimizes waste and reduces unnecessary expenses. This not only enhances surgeon, staff, and patient safety and satisfaction but also maximizes the utilization of operating room facilities, ultimately resulting in cost-effective care delivery3,4.

The introduction of femtosecond laser technology in cataract surgery offers promising advancements and precision in lens procedures. However, integrating this technology into existing workflows presents challenges in creating an efficient and cost-effective care structure. The incorporation of femtosecond laser requires careful evaluation and optimization of workflows to accommodate the added steps and equipment. By understanding the specific requirements and sequencing of tasks, surgeons can identify potential bottlenecks and implement changes that enhance efficiency and minimize disruption in the surgical process. Additionally, evaluating the cost-effectiveness of femtosecond laser usage, considering factors such as equipment costs, maintenance, and potential savings in overall patient care, is crucial for informed decision-making5-8.

Efficiency and cost-effectiveness are essential considerations in cataract surgery, given the increasing prevalence of cataracts and reductions in reimbursement rates. Understanding operating room workflows allows cataract surgeons to optimize processes, reduce delays, and achieve significant cost savings. Moreover, the integration of femtosecond laser technology in lens surgery necessitates careful evaluation and adaptation of workflows to ensure efficient utilization and seamless integration. By prioritizing efficiency, time savings, and cost reduction through workflow optimization and the adoption of innovative technologies, cataract surgeons can provide optimal patient care while addressing the challenges posed by evolving healthcare demands and financial constraints.

The objective of this study is to identify workflows that enhance surgical efficiency and enhance satisfaction among patients, surgeons, and staff by closely monitoring the timing and movements of patients, staff, and surgeons throughout their surgical journey. By analyzing the collected data, workflow efficiencies and best practices to optimize the surgical process can be identified.

ELIGIBILITY:
Inclusion Criteria:

* Subject (male or female) must be at least 21 years of age
* Subject must have had an operable cataract in the study eye
* Eligible for femtosecond laser treatment and phacoemulsification
* Subject elected to undergo cataract extraction

Exclusion Criteria:

• Subjects who have difficulty lying flat for a 1-hour time period (e.g., spinal stenosis, cervical neck injury, claustrophobia, anxiety disorder, etc.).

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects who have undergone previous cataract surgery and meet the inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2023-06-09 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2024-06-29 (Actual)

PRIMARY OUTCOMES:
Identification of the amount of time in seconds required to perform surgical actions relevant to the FLACS procedure | On day of surgery (Day 0), from beginning to end of surgical procedure
  Total seconds required for each step of the surgical procedure
Measurement of time in seconds that a patient is interacting with the surgical staff | On day of surgery, (Day 0), time in seconds from arrival in pre-op area to discharge from post-op area
  Time in seconds from arrival in pre-op area to discharge from post-op area
Amount of time in seconds required to prepare patient for surgery | On day of surgery, (Day 0), from beginning of patient interaction with staff until surgical procedure begins
  Amount of time in seconds that patient is present with surgical staff prior to surgical procedure

CONTACTS AND LOCATIONS:
Locations (1):
- North Georgia Eye Associates, Gainesville, Georgia, United States

IPD SHARING:
Plan to Share IPD: Undecided